CLINICAL TRIAL: NCT00038337
Title: Improving Functional Health Literacy in Older Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: E2569R
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-05

CONDITIONS: Visual And Cognitive Disability
Keywords: Health Literacy; Visual; Cognitive
MeSH Terms: interventions — Health Literacy

INTERVENTIONS:
Procedure: Health Literacy

SUMMARY:
The objective of this two parallel component study is to develop interventions for the visual and cognitive related health literacy disabilities of older veterans. The first component will test two interventions for improving functional health literacy performance (enhancing the design of health literacy materials and training reading skills) by using a 2 x 2 between subjects factorial design. The second component consists of patient, family, and provider focus groups who will help determine where to apply and disseminate the interventions by identifying problematic sources of text-based health materials. Finally, as a result of both components improved health information design guidelines and training protocols will be developed as rehabilitative interventions for health literacy disability.

DETAILED DESCRIPTION:
Objective of this two parallel component study is to develop interventions for the visual and cognitive related health literacy disabilities of older veterans. The first component will test two interventions for improving functional health literacy performance (enhancing the design of health literacy materials and training reading skills) by using a 2 x 2 between subjects factorial design. The second component consists of patient, family, and provider focus groups who will help determine where to apply and disseminate the interventions by identifying problematic sources of text-based health materials. Finally, as a result of both components, improved health information design guidelines and training protocols will be developed as rehabilitative interventions for health literacy disability.

Specific research questions are:

1. Can the lower functional health literacy performance of veterans be improved by following text design directives intended to account for age-related visual and cognitive changes (enhanced version)?
2. Does instruction in skills and strategies for reading yield improvements in functional health literacy performance?
3. Does instruction in reading skills and enhanced text design improve functional health literacy to a greater extent than either intervention alone?
4. Are reading gains maintained over time?
5. What everyday sources of functional health literature are problematic for today's veterans?
6. How do visual, cognitive, and descriptive factors contribute to change in functional health literacy score?
7. What is the functional health literacy of older veterans who utilize Atlanta VA health care?

Focus Groups: Three two-hour focus groups will be composed of 15 VA health professionals, 15 outpatient veterans aged 65 and older with low functional health literacy, and 15 family members of veterans with low functional health literacy. These focus groups will identify sources of text-based health information which they find to be problematic from their respective perspectives. These sources, as well as recommendations for the application and dissemination of guidelines and directives for improved health information designs and training protocols, will be compiled using transcription and analysis of focus group sessions.

Interventions: Community dwelling veterans aged 65 and older will be recruited from the Geriatric Primary Care Clinic and the Veteran's Learning Center. Ethnicity, education, health status, general literacy, and other descriptive information will be recorded. Visual baseline measures will include assessments of visual skills for reading and visual function. Cognitive baseline measures will include assessments of word recognition, text comprehension ability, verbal working memory, perceptual speed and vocabulary level. Functional health literacy, measured by the TOFHLA, will be the main outcome measure. This objective and standardized instrument measures the ability of adults to read and understand medical instructional and health care information presented in prose passages and passages containing numerical information. Two hundred and forty participants demonstrating inadequate functional health literacy scores (by the screening instrument STOFHLA) will be randomly assigned to one of four groups: control (N=60), enhanced only (N=60), reading skills and strategies instruction only (N=60), or enhanced with reading skills and strategies instruction (N=60). All participants will receive vision and cognition testing and will then participate in two 2-hour sessions. Depending on group assignment participants will either 1) read standard health-related material (control) 2) read enhanced health-related material (enhanced) 3) receive reading skills training (training) 4) receive reading skills training with enhanced materials (training and enhanced).

ELIGIBILITY:
Older Veterans

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2001-04; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D. Special Assistant to the Director — Program Analysis and Review Section (PARS), VA Rehabilitation Research & Development Service; Vicki Mongiardo, Program Analyst — Program Analysis and Review Section (PARS), VA Rehabilitation Research and Development Service
Locations (1):
- VA Medical Center, Decatur, Georgia, United States